CLINICAL TRIAL: NCT01090661
Title: A Randomized Double-Blinded Crossover Trial to Define the ECG Effects of Mipomersen (ISIS 301012) Using a Therapeutic and Supratherapeutic Dose Compared to Placebo and Moxifloxacin (a Positive Control) in Healthy Men and Women: A Thorough ECG Trial
Brief Title: A Study to Evaluate the Effect of Mipomersen on Cardiac Repolarization Conducted in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIPO2800209
Record Dates: First submitted 2010-03-18; First posted 2010-03-22 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: antisense; ApoB (Apolipoprotein B); LDL (low density lipoprotein); thorough QT
MeSH Terms: interventions — mipomersen; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- mipomersen IV (supra-therapeutic dose) (Experimental): 200 mg of mipomersen IV / placebo SC
  Interventions: Drug: mipomersen sodium; Drug: placebo
- mipomersen SC (therapeutic dose) (Experimental): 200 mg of mipomersen SC / placebo IV
  Interventions: Drug: mipomersen sodium; Drug: placebo
- moxifloxacin IV (Active Comparator): 400 mg of moxifloxacin IV / placebo SC
  Interventions: Drug: moxifloxacin hydrochloride (Avelox®); Drug: placebo
- placebo (Placebo Comparator): Placebo IV / placebo SC
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: mipomersen sodium — 200 mg of mipomersen intravenous (IV) (single dose)
  Other Names: ISIS 301012
  Arms: mipomersen IV (supra-therapeutic dose)
Drug: mipomersen sodium — 200 mg of mipomersen subcutaneous (SC) (single dose)
  Other Names: ISIS 301012
  Arms: mipomersen SC (therapeutic dose)
Drug: moxifloxacin hydrochloride (Avelox®) — 400 mg of moxifloxacin intravenous (IV) single dose
  Arms: moxifloxacin IV
Drug: placebo — placebo intravenous (IV) single dose
  Arms: mipomersen SC (therapeutic dose); placebo
Drug: placebo — placebo subcutaneous (SC) single dose
  Arms: mipomersen IV (supra-therapeutic dose); moxifloxacin IV; placebo

SUMMARY:
To assess the electrocardiogram (ECG) effects of mipomersen administered as a 200-mg subcutaneous (SC) therapeutic and a 200-mg intravenous (IV; [2-hour infusion]) supra-therapeutic dose relative to placebo in healthy adult male and female subjects; and to evaluate the safety and pharmacokinetics (PK) of mipomersen when administered as a single therapeutic (200 mg) SC and a single, supra-therapeutic (200 mg) IV dose.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, single-site, crossover study in healthy male and female subjects to determine if mipomersen administered as a single therapeutic (200 mg) SC and a single supra-therapeutic (200 mg) IV dose delays cardiac repolarization as determined by the measurement of QT/corrected QT (QTc) interval. A total of 60 healthy male and female subjects will be enrolled in this 4-way crossover study, randomly assigned to 1 of 8 treatment sequences, and cross over into 4 treatment periods where each subject will receive both a single SC injection and a single IV infusion during each period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided before any study-related procedures are performed.
* Body mass index (BMI) of 19 to 32 kg/m2 inclusive.
* Subjects can not have consumed nicotine or nicotine-containing products for at least 6 months before Screening.
* Subjects are nonpregnant and nonlactating, surgically sterile, postmenopausal, abstinent, or subject or partner is willing to use a reliable method of contraception during the study and 5 months after the last dose of investigational product.

Exclusion Criteria:

* History of risk factors for Torsades de Pointes, known Long QT Syndrome, heart failure, myocardial infarction, angina, or clinically significant abnormal laboratory assessments or family history of Long QT or Brugada Syndrome.
* Abnormal screening ECG that is interpreted by the Investigator to be clinically significant.
* Use of concomitant medications (prescribed or over-the-counter), without the approval of the Investigator and Sponsor, within 7 days before the first dose of investigational product.
* Clinically significant abnormal findings on the physical examination, ECG, blood pressure, heart rate, medical history, or clinical laboratory results at Screening or before dosing.
* History of clinically significant allergies or hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease.
* Positive test for HIV antibody, hepatitis C antibody, or hepatitis B surface antigen.
* Positive test for drugs of abuse, alcohol, or cotinine at Screening or before dosing or history of drug or alcohol abuse or dependence within 1 year before Screening.
* History of cancer, with the exception of basal cell carcinoma.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
change from baseline in QTcF (corrected Frederica's CT interval) | ECG monitoring up to 24 hours post dose

SECONDARY OUTCOMES:
ECG intervals (QTcB (corrected Bazett's QT interval), HR (heart rate, PR, QRS, and QT) | ECG monitoring up to 24 hours post dose
change in ECG morphological patterns | ECG monitoring up to 24 hours post dose
Correlation between delta delta QTc interval and plasma mipomersen concentrations | ECG monitoring up to 24 hours post dose
Incidence of treatment-emergent Adverse Events | Assessed at each visit
mipomersen plasma pharmacokinetic (PK) parameters: Area Under the Curve (AUC 0-22.5h), Maximum Concentration (Cmax), Time to Maximum Concentration (Tmax) | Serial PK sampling up to 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- PPD Development, LP, Austin, Texas, United States